CLINICAL TRIAL: NCT04240093
Title: CoMBAT Opioid Use Disorder: A Pilot Randomized Controlled Trial of a Combined Medication and Behavioral Activation Treatment for People Living With Opioid Use Disorder
Brief Title: CoMBAT Opioid Use Disorder: A Combined Medication and Behavioral Activation Treatment for People Living With Opioid Use Disorder
Acronym: CoMBAT_OUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Boston University (Other); University of Massachusetts, Boston (Other); National Institute of General Medical Sciences (NIGMS) (NIH); Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1906002463; Junior Investigator Award (Other Grant/Funding Number: COBRE on Opioids and Overdose); 5P20GM125507-02 (NIH)
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Results first posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Opioid-use Disorder; Medication Adherence; Health Care Utilization
Keywords: Medications for opioid use disorder; Methadone; Buprenorphine; Behavioral Activation
MeSH Terms: conditions — Opioid-Related Disorders; Medication Adherence; Patient Acceptance of Health Care | interventions — Therapeutics; Dosage Forms

STUDY DESIGN:
Intervention Model Description: Two-arm RTC, randomized 1:1 to two arms: (1) the CoMBAT intervention (behavioral activation and substance abuse/health navigation) counseling, which lasts ten sessions; and (2) the standard of care comparison condition, including two equivalent substance abuse/ health navigation counseling sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental: Behavioral Activation (8 sessions) + Substance Abuse and Health Navigation Counseling (2 sessions) + Meds
  Interventions: Behavioral: Behavioral Activation (BA) Therapy; Behavioral: Substance Abuse and Health Navigation Counseling; Other: Medications for Opioid Use Disorder
- Standard of Care (Active Comparator): Substance Abuse and Health Navigation Counseling (2 sessions) + Meds
  Interventions: Behavioral: Substance Abuse and Health Navigation Counseling; Other: Medications for Opioid Use Disorder

INTERVENTIONS:
Behavioral: Behavioral Activation (BA) Therapy — 8 sessions of behavioral activation therapy
  Arms: Experimental
Behavioral: Substance Abuse and Health Navigation Counseling — 2 standard substance abuse and health navigation counseling
Other: Medications for Opioid Use Disorder — Medications for opioid use disorder (i.e., buprenorphine and methadone) as prescribed by a community provider (not provided as part of the study).

SUMMARY:
This study seeks primarily to test, in a two-arm randomized controlled trial (RCT), the feasibility, acceptability, and preliminary efficacy of CoMBAT OUD, an intervention that integrates Behavioral Activation (BA) and substance abuse and health navigation counseling for individuals who are receiving medications for opioid use disorder (i.e., methadone; suboxone) to help them improve engagement in care and opioid use treatment outcomes. Participants will be randomized 1:1 to two arms: (1) the CoMBAT intervention (2 sessions of substance abuse and health navigation counseling + 8 sessions of BA counseling); or the (3) the standard of care (SOC) comparison condition, including two equivalent substance abuse and health navigation counseling. Participants will be followed for 6 months post-randomization, with assessments at months 3 and 6.

DETAILED DESCRIPTION:
Opioid use disorder (OUD) is a chronic, relapsing disease and a major source of morbidity and mortality in the United States. Medications for opioid use disorder (i.e., methadone; buprenorphine) have been shown to reduce opioid use in diverse populations; however, long-term use of these medications and engagement in care are often suboptimal. Depression has been shown to contribute to medication discontinuation and care disengagement. Behavioral activation (BA) therapy is an evidence-based, behavioral treatment that has been shown to be effective in treating comorbid depression and substance use in diverse populations with smoking, alcohol, stimulant, and poly-substance use disorder. BA utilizes therapeutic techniques that help patients gradually increase goal-directed, potentially rewarding and pleasurable activities while decreasing the intensity and frequency of adverse events and consequences in order to improve mood. Given that BA utilizes strategies that can support individuals in alleviating depression and build the capacity to navigate life challenges, pairing BA with medications for OUD could help to ensure continued engagement in care and improve OUD treatment outcomes.

This study, therefore, seeks to determine the feasibility of study procedures, enhance participant acceptability, and demonstrate preliminary efficacy of the CoMBAT (Combined Medication and Behavioral Activation Treatment) intervention. The investigators will enroll individuals currently being treated with methadone or buprenorphine for OUD in a pilot randomized controlled trial (RCT) of the CoMBAT intervention. Prior to randomization, participants will receive 2 health navigation and standard substance abuse counseling sessions. Participants will then be equally randomized to either: 1) the 8-session CoMBAT intervention; or 2) standard of care. The primary outcome is engagement in care. Secondary outcomes include self-reported days of opioid use and opioid-positive urinalysis. Intervention feasibility and acceptability will also be assessed. Participants will complete major assessment visits (survey and toxicology testing) at baseline and 3- and 6-months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Initiated medications for opioid use >= 30 day prior to screening
* Current depressive symptoms
* Plans to stay in Rhode Island or Massachusetts for at least 6-months
* Able to read, speak, and understand English
* Willing and able to provide informed consent

Exclusion Criteria:

* Does not plan to continue taking medications for opioid use disorder
* Unable to provide informed consent due to severe mental or physical illness, or substance intoxication at the time of interview
* Discovery of active suicidal ideation at the time of interview
* In the second or third trimester of pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn W Hughto, PhD, MPH, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw data for additional analysis will be available to outside individuals through contacting the Principal Investigator (PI) at two different times. The first will be after all of the baseline data is collected. The PI will institute a concept plan process where internal study staff first have the availability to write papers or give presentations on particular topics. After this, if outside individuals wish to analyze the data, the PI will welcome this collaboration. A similar process will happen for outcome data; however, this will not be possible until the publication and release of the outcome paper(s). The PI will allow access for pooled data analysis projects, or projects for outside individuals. Information regarding the availability of data for analysis will be listed on the PIs' web page. Contact information for the PI will be listed in all manuscripts and publications as another means to access data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The first time point at which outside investigators may request IPD will be after all of the baseline data has been collected and internal study staff have been offered the availability to write papers or give presentations on particular topics. A similar process will take place for outcome data following publication and release of the outcome paper(s). The PI will store the data indefinitely.
Access Criteria: Raw data for additional analysis will be available to outside individuals by contacting the Principal Investigator (PI). The PI will institute a concept plan process where internal study staff first have the availability to write papers or give presentations on particular topics. After this, if outside individuals wish to analyze data, the PI will welcome this collaboration. The PI will allow access for pooled data analysis projects, or projects for outside individuals. Information regarding the availability of data for analysis will be listed on the PI's web page (see below).
URL: http://www.fresh-research.com

REFERENCES:
- See also: FRESH Research Lab — http://www.fresh-research.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via ads posted online (i.e., Craigslist) and in-person at outpatient substance use treatment clinics and community organizations serving people who use drugs in Rhode Island and Massachusetts. Substance use treatment providers and staff also provided direct referrals and snowball sampling was used.
Pre-assignment Details: A total of 44 individuals consented; of these, 12 individuals were lost to follow-up prior to randomization, resulting in a randomized sample of 32 participants (16 CoMBAT experimental arm; 16 Standard of Care control arm).
Period: Overall Study
Arm/Group | Experimental | Standard of Care
Started | 16 | 16
3 Month Follow-Up | 14 | 16
6 Month Follow Up | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for all enrolled and randomized participants (n=32).
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Standard of Care | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (10.98) | 39.4 (11.6) | 39.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 8 | 13 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 16 | 13 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  White | 12 | 13 | 25
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Medication Type [Count of Participants; unit: Participants]
  Methadone | 12 | 11 | 23
  Buprenorphine | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Missed Medication Doses - Past 30 Days
Description: Self-reported change in the number of missed methadone or buprenorphine doses in the past 30 days. Raw, unadjusted means at 6-month follow-up are reported.
Time Frame: Baseline, 3 month follow-up, and 6 month follow-up
Population: Intent to Treat Analysis. For the unadjusted means by time-point data, there were missing data for 2 participants in the CoMBAT experimental arm at the 3-month follow-up visit.
Measure: Mean (Standard Deviation); unit: Number of missed doses
Groups:
- CoMBAT (Experimental): Experimental: Behavioral Activation (8 sessions) + Substance Abuse and Health Navigation Counseling (2 sessions) + Meds
  Behavioral Activation (BA) Therapy: 8 sessions of behavioral activation therapy
  Substance Abuse and Health Navigation Counseling: 2 standard substance abuse and health navigation counseling
  Medications for Opioid Use Disorder: Medications for opioid use disorder (i.e., buprenorphine and methadone) as prescribed by a community provider (not provided as part of the study).
- Standard of Care (SOC; Control): Substance Abuse and Health Navigation Counseling (2 sessions) + Meds
  Substance Abuse and Health Navigation Counseling: 2 standard substance abuse and health navigation counseling
  Medications for Opioid Use Disorder: Medications for opioid use disorder (i.e., buprenorphine and methadone) as prescribed by a community provider (not provided as part of the study).
Arm/Group | CoMBAT (Experimental) | Standard of Care (SOC; Control)
Number analyzed (Participants) | 16 | 16
Number of missed doses
  Baseline | 3.13 (3.48) | 2.81 (3.00)
  3 Month Follow-Up: number analyzed (Participants) | 14 | 16
  3 Month Follow-Up | 3.71 (4.41) | 2.25 (3.00)
  6 Month Follow-Up | 1.19 (2.43) | 1.69 (4.29)
Statistical Analysis 1: Comparison: CoMBAT (Experimental) vs Standard of Care (SOC; Control); Hypothesis: The CoMBAT intervention arm would be superior to the Standard of Care control arm with regard to reductions in missed medication doses in the past 30 days at follow-up; Test type: Superiority — This is a pilot intervention trial and was not powered to detect statistical significance; p = 0.17, Generalized estimating equations (GEE) — a priori alpha p<0.05; Generalized estimating equations (GEE) with a poisson distribution controlling for baseline values; Beta coefficient = -0.46, 95% CI 2-sided [-1.11 to 0.20], Standard Error of Mean 0.33

2. Primary Outcome: Number of Missed Medication-related Visits - Past 30 Days
Description: Self-reported change in the number of medication-related clinic visits missed in the past 30 days from baseline to follow-up.
Time Frame: Baseline, 3 month follow-up, and 6 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of missed visits
Arm/Group | CoMBAT (Experimental) | Standard of Care (SOC; Control)
Number analyzed (Participants) | 16 | 16
Number of missed visits
  Baseline | 1.13 (1.20) | 0.94 (0.85)
  3 Month Follow-Up: number analyzed (Participants) | 14 | 16
  3 Month Follow-Up | 0.14 (0.36) | 0.25 (0.45)
  6 Month Follow-Up | 0.06 (0.03) | 0.06 (0.35)
Statistical Analysis 1: Comparison: CoMBAT (Experimental) vs Standard of Care (SOC; Control); Hypothesis: The CoMBAT intervention arm would be superior to the Standard of Care control arm with regard to reductions in missed medication-related visits in the past 30 days at follow-up; Test type: Superiority — This pilot feasibility and acceptability study was not powered to detect a statistically significant effect; p = 0.90, Generalized estimating equation (GEE) — a priori alpha p<0.05; Generalized estimating equations (GEE) with a Poisson distribution controlling for baseline values; Beta coefficient = -0.18, 95% CI 2-sided [-3.09 to 2.72], Standard Error of Mean 1.48

3. Secondary Outcome: Fentanyl and Opiate-positive Urine Toxicology Screen
Description: Fentanyl or opiate-positive urine screen (opiates refer to natural opioids such as heroin, morphine so buprenorphine, methadone, and other synthetic opioids are not included)
Time Frame: Baseline, 3 month follow-up, and 6 month follow-up
Population: Intent to Treat Analysis. For the raw count data, there were missing data for 2 participants in the CoMBAT experimental arm at the 3-month follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | CoMBAT (Experimental) | Standard of Care (SOC; Control)
Number analyzed (Participants) | 16 | 16
Participants
  Baseline | 6 | 3
  3 Month Follow-Up: number analyzed (Participants) | 14 | 16
  3 Month Follow-Up | 3 | 4
  6 Month Follow-Up | 2 | 3
Statistical Analysis 1: Comparison: CoMBAT (Experimental) vs Standard of Care (SOC; Control); Hypothesis: Fewer participants in the CoMBAT experimental arm will have a positive opioid toxicology screen at the 6-month follow-up compared to participants in the SOC control arm; Test type: Superiority — As a pilot feasibility and acceptability trial, this study was not powered to detect a statistically significant effect; p = 0.02, Generalized estimating equations (GEE) — A priori alpha p<0.05; Generalized estimating equation (GEE) modeling with a binomial distribution, controlling for baseline values; Beta coefficient = -4.71, 95% CI 2-sided [-8.72 to -0.70], Standard Error of Mean 2.05

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Experimental | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-03-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT04240093/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT04240093/SAP_002.pdf
  • Informed Consent Form (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT04240093/ICF_001.pdf